CLINICAL TRIAL: NCT02972957
Title: A Study of Intranasal Live Attenuated Influenza Vaccine Immunogenicity and Associations With the Nasopharyngeal Microbiome Among Children in the Gambia - The NASIMMUNE Study
Brief Title: A Study of Intranasal Live Attenuated Influenza Vaccine Immunogenicity and Associations With the Nasopharyngeal Microbiome Among Children in the Gambia
Acronym: NASIMMUNE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: University of Edinburgh (Other); Public Health England (Other Government); University of Oxford (Other); National Institute for Public Health and the Environment (RIVM) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SCC 1502
Record Dates: First submitted 2016-11-17; First posted 2016-11-25 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Influenza
Keywords: intranasal; flu vaccine; Gambian children
MeSH Terms: conditions — Influenza, Human | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- LAIV-vaccinated group 1 (Experimental): Nasovac-S vaccination group A , blood samples days 0, 2, 21
  Interventions: Biological: Nasovac-S
- LAIV-vaccinated group 2 (Experimental): Nasovac-S vaccination group B, blood samples at days 0, 7, 21
  Interventions: Biological: Nasovac-S
- Unvaccinated (No Intervention): control group C
- Oral Azithromycin & vaccination (Experimental): group D - a single dose of oral Azithromycin will be given 28 days prior to Nasovac-S vaccination
  Interventions: Biological: Nasovac-S; Drug: Azithromycin

INTERVENTIONS:
Biological: Nasovac-S — one of 0.5ml intranasal dose of trivalent live attenuated vaccine (LAIV)
  Arms: LAIV-vaccinated group 1; LAIV-vaccinated group 2; Oral Azithromycin & vaccination
Drug: Azithromycin — a single dose of Azithromycin (liquid formulation - Zithromax) at 20mg/Kg (up to a maximum adult dose 1g) to be given to a subset of subjects
  Other Names: Zithromax
  Arms: Oral Azithromycin & vaccination

SUMMARY:
The live attenuated influenza vaccine (LAIV) is made up of weakened influenza viruses given into the nose and in early studies was shown to be better than the standard influenza vaccine at preventing infections in children. However, more recently, it has performed less well and it may also work less well in Sub-Saharan Africa. Not only do the investigators not know why this is, but the investigators also do not fully understand why LAIV produces stronger nasal antibody responses in some individuals but not others. Usually harmless bacteria that are present in participants noses can influence how our immune system works and variations in these may explain differences in how LAIV works. The project will recruit children given LAIV in the Gambia to gain further understanding of these issues.

The investigators will measure a variety of responses to LAIV, including genes that can change their expression early after vaccination and use advanced computational techniques to identify new relationships between these genes and other LAIV responses. The investigators will also see whether nasal bacterial profiles in children who respond to LAIV are different from those who do not. In addition, the investigators will alter these bacteria in a subset of children with antibiotics and see whether this affects both nasal gene expression and later responses to LAIV.

DETAILED DESCRIPTION:
Purpose The overall goal of this study is to conduct at detailed immunogenicity study of intranasal live attenuated influenza vaccine (LAIV; Nasovac-S, Serum Institute of India Pvt. Ltd.), including identification of early molecular signatures associated with a robust mucosal immune response. In addition, the study team will explore whether the nasopharyngeal microbiome influences this immune response and whether LAIV has an impact on the microbiome.

A total of 365 healthy children aged 24 - 59 months will be recruited in The Gambia for this study.

Background Both the burden of infection and use of influenza vaccines in children from sub-Saharan Africa (SSA) have been neglected. There are limited immunogenicity or efficacy data from SSA of the widely used Ann Arbor strain-derived LAIV. This LAIV was shown to have greater relative efficacy compared to inactivated influenza vaccine in children in early randomized-controlled trials. There has, however, been concern regarding lower vaccine effectiveness in the US in recent years.

The Serum Institute of India Pvt. Ltd. has recently developed a trivalent LAIV (Nasovac-S) via a WHO facilitated donation of a Russian-derived LAIV, with the intention of scaling up provision of LAIV to resource-limited settings. Based on initial safety and immunogenicity data, Nasovac-S was licensed in India and granted a WHO prequalification certificate in 2015. Two placebo-controlled efficacy studies using Nasovac-S were recently undertaken in Bangladesh and Senegal (in children aged 24 - 59 months and 24 - 71 months respectively), providing mixed and contrasting results. In Senegal, no efficacy was found against the circulating pandemic H1N1 influenza strain (-9.7%, 95% CI -62.6, 26.1). In Bangladesh the overall vaccine efficacy to vaccine-matched strains, in a study of identical design, was 57.5% (95% CI 43.6, 68.0), with efficacy against H1N1 and H3N2, 50.0% (95% CI 9.2, 72.5) and 60.4% (95% CI 44.8, 71.6) respectively. The reason for the discrepancy in these studies or the poorer performance of the H1N1 component is not clear and emphasizes the need to undertake detailed immunogenicity studies of this vaccine in SSA. On a wider note, the exact immunological mechanisms of action of LAIV are also under-explored.

Study type:

Interventional

Design:

All primary objectives will be addressed through the conduct of a phase 4, randomized, controlled clinical vaccine trial. A total of 330 healthy children aged 24 - 59 months will be enrolled into one of three groups of equal size (3 x 110 children):

(i) LAIV-vaccinated (Group A - blood sample at day 0, 2, 21) (ii) LAIV-vaccinated (Group B - blood sample at day 0, 7, 21) (iii) Control group (Group C)

The study is not blinded, but group allocation will be concealed from the investigator team and block randomization stratified by sex will be undertaken.

Two LAIV-vaccinated groups are included in order to achieve several exploratory objectives, which require blood sampling at different times following vaccination, whilst minimizing the number of times children are bled. The unvaccinated subjects will serve as a control group for the primary objective of assessing the impact of LAIV on the nasopharyngeal microbiome.

An additional 35 healthy children aged 24 - 59 months will be recruited in the 2nd phase of recruitment (approximately Jan - June 2018) to assess how modulation of the nasopharyngeal microbiome with antibiotics impacts the mucosal immunogenicity to LAIV. These subjects will be matched as closely as possible by pre-antibiotic nasopharyngeal microbiome profile, age and sex (in that order of preference), in an exploratory nested case-control study, to n = 35 children recruited in the main clinical trial.

Official title A Study of Intranasal Live Attenuated Influenza Vaccine Immunogenicity and Associations with the Nasopharyngeal Microbiome Among Children in the Gambia (The NASIMMUNE study)

Primary outcome measures

* To identify novel early systemic and mucosal molecular signatures following LAIV that are associated with subsequent robust nasal and oral influenza-specific immunoglobulin A (IgA) responses, in order to provide insight into the mechanisms of successful mucosal immunization
* To identify associations between nasopharyngeal microbiota and nasal and oral influenza-specific IgA responses post-LAIV in Gambian children, to explore whether microbiome variability can explain suboptimal immune responses in some individuals to live intranasal mucosal vaccines in Sub-Saharan Africa
* To establish whether LAIV impacts the nasopharyngeal microbiome, with a specific focus on the burden of S. pneumoniae

ELIGIBILITY:
Inclusion Criteria:

* • Healthy male or female child at least 24 months of age and less than 60 months of age at the time of study entry.

  * Resident in the study area and with no plans to travel outside the study area during the period of subject participation.
  * Informed consent for the study participation obtained from a parent (or guardian only if neither parent is alive or if guardianship has been legally transferred (see section 11.2).
  * Willingness and capacity to comply with the study protocol as judged by a member of the clinical trial team.

Exclusion Criteria:

* • Serious, active, medical condition, including but not limited to:

  * chronic disease of any body system
  * severe protein-energy malnutrition (weight-for-height Z-score of less than -3)
  * known genetic disorders, such as Down's syndrome or other cytogenetic disorder

    * Active wheezing
    * History of documented hypersensitivity to eggs or other components of the vaccine (including gelatin, sorbitol, lactalbumin and chicken protein), or with life-threatening reactions to previous influenza vaccinations.
    * History of documented hypersensitivity to macrolide antibiotics
    * History of Guillain-Barré syndrome.
    * Receipt of aspirin therapy or aspirin-containing therapy within the two weeks before planned study vaccination.
    * Any suspected or confirmed congenital or acquired state of immune deficiency including but not limited to primary immunodeficiencies including thymus disorders, HIV/AIDS, hematological or lymphoid malignancies (blood tests will not be routinely undertaken with this regard as part of the study).
    * Any current immunosuppressive/immunomodulatory treatment or receipt of any such treatment within the six months preceding trial enrolment (for corticosteroids this is defined as a dose of prednisolone (or equivalent) of greater than 2mg/kg/day for one week or 1mg/kg/day for one month. The use of topical corticosteroids is not an exclusion criterion.
    * The use of inhaled corticosteroids within the last one month.
    * Receipt of an influenza vaccine within the past 12 months.
    * Has any condition determined by investigator as likely to interfere with evaluation of the vaccine or be a significant potential health risk to the child or make it unlikely that the child would complete the study.
    * Any significant signs or symptoms of an acute illness or infection including:
  * an axillary temperature of 38.0°C or above or documented fever of 38°C or above in the preceding 14 days.
  * Any acute respiratory infection within 14 days of enrollment visit. If the reason for ineligibility is likely to be temporary (e.g. a fever of 38°C or above or acute respiratory infection) and either will or may resolve before the infant reaches 60 months, they will not be recorded as a screening failure but instead will be re-screened within an appropriate future time-window (e.g. at least 14 days after the last documented fever of 38°C or above or resolution of respiratory illness) and a decision made regarding eligibility at that point.

Ages: 24 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 364 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2019-05-23 (Actual)

PRIMARY OUTCOMES:
nasal IgA response | 21 days post LAIV
  Influenza specific nasal IgA responses
fold increase in oral fluid influenza-specific/total IgA ratio | day 0 - Day 21
fold increase in oral fluid influenza-specific/total IgG ratio | Day 0 - Day 21

SECONDARY OUTCOMES:
density of S. Pneumoniae | day 7 and day 21 after LAIV compared to day 0
  density of S. Pneumoniae before and after LAIV as established by quantitative PCR
Changes in the relative abundance of different operational taxanomic units (OTUs) of nasopharyngeal microbiota | day 7 and day 21 compared to day 0 in each participant
gene expression changes in nasal and systemic samples | 2 days after LAIV

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Research Council unit The Gambia, Banjul, The Gambia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peno C, Jagne YJ, Clerc M, Balcazar Lopez C, Armitage EP, Sallah H, Drammeh S, Senghore E, Goderski G, van Tol S, Meijer A, Ruiz-Rodriguez A, de Steenhuijsen Piters WAA, de Koff E, Jarju S, Lindsey BB, Camara J, Bah S, Mohammed NI, Kampmann B, Clarke E, Dockrell DH, de Silva TI, Bogaert D. Interactions between live attenuated influenza vaccine and nasopharyngeal microbiota among children aged 24-59 months in The Gambia: a phase 4, open-label, randomised controlled trial. Lancet Microbe. 2025 Mar;6(3):100971. doi: 10.1016/j.lanmic.2024.100971. Epub 2025 Jan 17. PMID 39832517
- [Derived] Keeley AJ, Groves D, Armitage EP, Senghore E, Jagne YJ, Sallah HJ, Drammeh S, Angyal A, Hornsby H, de Crombrugghe G, Smeesters PR, Rossi O, Carducci M, Peno C, Bogaert D, Kampmann B, Marks M, Shaw HA, Turner CR, de Silva TI. Streptococcus pyogenes Colonization in Children Aged 24-59 Months in the Gambia: Impact of Live Attenuated Influenza Vaccine and Associated Serological Responses. J Infect Dis. 2023 Oct 3;228(7):957-965. doi: 10.1093/infdis/jiad153. PMID 37246259
- [Derived] Peno C, Armitage EP, Clerc M, Balcazar Lopez C, Jagne YJ, Drammeh S, Jarju S, Sallah H, Senghore E, Lindsey BB, Camara J, Bah S, Mohammed NI, Dockrell DH, Kampmann B, Clarke E, Bogaert D, de Silva TI. The effect of live attenuated influenza vaccine on pneumococcal colonisation densities among children aged 24-59 months in The Gambia: a phase 4, open label, randomised, controlled trial. Lancet Microbe. 2021 Dec;2(12):e656-e665. doi: 10.1016/S2666-5247(21)00179-8. PMID 34881370
- [Derived] Lindsey BB, Jagne YJ, Armitage EP, Singanayagam A, Sallah HJ, Drammeh S, Senghore E, Mohammed NI, Jeffries D, Hoschler K, Tregoning JS, Meijer A, Clarke E, Dong T, Barclay W, Kampmann B, de Silva TI. Effect of a Russian-backbone live-attenuated influenza vaccine with an updated pandemic H1N1 strain on shedding and immunogenicity among children in The Gambia: an open-label, observational, phase 4 study. Lancet Respir Med. 2019 Aug;7(8):665-676. doi: 10.1016/S2213-2600(19)30086-4. Epub 2019 Jun 21. PMID 31235405
- [Derived] Armitage EP, Camara J, Bah S, Forster AS, Clarke E, Kampmann B, de Silva TI. Acceptability of intranasal live attenuated influenza vaccine, influenza knowledge and vaccine intent in The Gambia. Vaccine. 2018 Mar 20;36(13):1772-1780. doi: 10.1016/j.vaccine.2018.02.037. Epub 2018 Feb 23. PMID 29483030